CLINICAL TRIAL: NCT02128360
Title: Analysis of IVF Outcome After Minimal Stimulation vs. High Dose Stimulation for Patients With Low Ovarian Reserve
Brief Title: Comparison of 2 Ovarian Stimulation Protocols for Women With Low Ovarian Reserve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-14-1034-SD-CTIL
Record Dates: First submitted 2014-03-23; First posted 2014-05-01 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Infertility
Keywords: Low ovarian reserve; Poor responder; Infertility
MeSH Terms: conditions — Infertility | interventions — Letrozole; Gonadotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minimal stimulation protocol (Active Comparator): Low dose Letrozole 2.5 mg over 5 days, starting from cycle day 2, overlapping with low dose gonadotropins, starting from day 3 of the Letrozole at 150 units per day. GnRH antagonist to avoid premature LH surge will be introduced when one or more of the growing follicles reached approximately 14 mm in size
  Interventions: Drug: Letrozole, Gonadotropins
- High dose protocol (Active Comparator): High dose of gonadotropins (≥300 IU/day) starting from cycle day 3. GnRH antagonist will be introduced to avoid premature LH surge when one or more of the growing follicles will reach approximately 14 mm in size
  Interventions: Drug: Gonadotropins

INTERVENTIONS:
Drug: Letrozole, Gonadotropins
  Arms: Minimal stimulation protocol
Drug: Gonadotropins
  Arms: High dose protocol

SUMMARY:
The purpose of this study is to determine whether minimal ovarian stimulation for in vitro fertilization is superior to high dose stimulation. Number of mature eggs, number of embryos as well as pregnancy rates will be compared.

DETAILED DESCRIPTION:
A prospective randomized trial will be carried out. The Minimal stimulation (MS) protocol is based on low dose letrozole 2.5 mg over 5 days, starting from cycle day 2, overlapping with low dose gonadotropins, starting from day 3 of the letrozole at 150 units per day. GnRH antagonist wil be introduced to avoid premature LH surge when one or more of the growing follicles reached approximately 14 mm in size. The high dose stimulation protocol is based on high dose of gonadotropins (≥300 IU/day) throughout the cycle with the usage of gonadotropin-releasing hormone (GnRH) antagonist to avoid premature luteinizing hormone (LH) surge as described above.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of poor responder to ovarian stimulation

Exclusion Criteria:

* Patients undergoing pregestational diagnosis (PGD)
* Patients using donor eggs

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rates | 1 Year

SECONDARY OUTCOMES:
Number of High quality embryos | 1 year
  How many embryos of 6-8 cells with low fragmentation in each arm
Number of eggs retrieved | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shir Dar, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- The Chaim Sheba Medical Center, Tel Litwinsky, Israel